CLINICAL TRIAL: NCT03669068
Title: Gastrointestinal Endoscopy in Patients With Prothrombotic Conditions: A Prospective, Multicentre, and Observational Registry
Brief Title: Gastrointestinal Endoscopy in Patients With Prothrombotic Conditions: THE ENDOHEM REGISTRY
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Collaborators: University of Salamanca (Other); Hospital Universitario Central de Asturias (Other); Hospital Universitario 12 de Octubre (Other); Puerta de Hierro University Hospital (Other); Hospital del Mar (Other); Hospital de Viladecans (Other); Hospital Clinic of Barcelona (Other); Hospital de Avilés (Unknown); Hospital General de Villalba (Unknown); Hospital General de Granollers (Unknown); Hospital Sant Pau (Unknown)
Responsible Party: Principal Investigator, Enrique Rodríguez de Santiago, Principal Investigator. MSc. Gastroenterologist, Hospital Universitario Ramon y Cajal
Other Study IDs: HRC-ENDOHEM-02
Record Dates: First submitted 2018-09-08; First posted 2018-09-13 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Gastrointestinal Bleeding; Cardiovascular Complication; Anticoagulants; Circulating, Hemorrhagic Disorder; Gastrointestinal Endoscopy
Keywords: Gastrointestinal endoscopy; Oral anticoagulants; Gastrointestinal bleeding; Cardiovascular event
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Hemorrhagic Disorders | interventions — Endoscopy, Gastrointestinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Elective endoscopy: Patients undergoing gastrointestinal endoscopy unrelated to anticoagulant-induced gastrointestinal bleeding.
  Interventions: Procedure: Gastrointestinal endoscopy
- Gastrointestinal bleeding: Patients with anticoagulant-induced gastrointestinal bleeding will be analyzed separately
  Interventions: Procedure: Gastrointestinal endoscopy

INTERVENTIONS:
Procedure: Gastrointestinal endoscopy — Two separated groups will be included in the registry:
  1. Patients with oral anticoagulants-induced gastrointestinal bleeding unrelated to an endoscopic procedure.
  2. Patients undergoing elective gastrointestinal endoscopy.

SUMMARY:
This observational study evaluates the safety of gastrointestinal endoscopy in patients on oral anticoagulants (Vitamin K antagonists, rivaroxaban, dabigatran, edoxaban, and apixaban). This registry aims to assess the incidence, characteristics and risk factors for cardiovascular and bleeding events associated with an endoscopic procedure. Besides, it aims to evaluate the differences between Vitamin K antagonists and DOACs users and to estimate the impact of anticoagulation withdrawal time on the primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years.
* Patients with preoperative use of oral anticoagulants (Vitamin K antagonist, apixaban, edoxaban, rivaroxaban or dabigatrán) undergoing gastrointestinal endoscopy.
* Patients on oral anticoagulants (Vitamin K antagonist, apixaban, edoxaban, rivaroxaban or dabigatran) presenting with gastrointestinal bleeding, regardless of receiving gastrointestinal endoscopy.
* Signed informed consent.

Exclusion Criteria:

* Negative to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on oral anticoagulants (Vitamin K antagonist, apixaban, edoxaban, rivaroxaban or dabigatran)
Sampling Method: Non-Probability Sample
Enrollment: 1602 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Cardiovascular events | 3 months
  Nº of patients during the study period presenting with a cardiovascular event, defined as any of the following entities: pulmonary thromboembolism, venous thromboembolism, acute coronary syndrome, arterial peripheral embolism or cerebrovascular accident.

SECONDARY OUTCOMES:
Incidence of therapeutic endoscopy-related gastrointestinal bleeding | 3 months
  Nº of patients during the study period presenting with therapeutic endoscopy-related gastrointestinal bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Available. Timeframe: 2018-2021
Access Criteria: Accredited researchers. The protocol is available in Spanish and will be provided by contacting the principal investigator.